CLINICAL TRIAL: NCT05186597
Title: Incidence of Multisystem Inflammatory Syndrome in Children (MIS-C) and Other Complications Following SARS-CoV-2. A Nationwide Population-based Study.
Brief Title: Incidence of MIS-C and Other Complications Following SARS-CoV-2 Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Innovation Fund Denmark (Individual); Ministry of Education, Denmark (Other Government)
Responsible Party: Principal Investigator, Ulrikka Nygaard, Primary investigator, Rigshospitalet, Denmark
Other Study IDs: H-20028631_MIS-C
Record Dates: First submitted 2022-01-09; First posted 2022-01-11 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: SARS CoV 2 Infection; Multisystem Inflammatory Disease, Pediatric, COVID-19 Related; Multisystem Inflammatory Syndrome in Children; COVID-19 Pandemic
Keywords: SARS CoV 2 Infection; Multisystem Inflammatory Syndrome in Children; COVID-19 Pandemic
MeSH Terms: conditions — COVID-19; pediatric multisystem inflammatory disease, COVID-19 related

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Multisystem inflammatory syndrome in children (MIS-C) is a rare severe complication to SARS-CoV-2 infection in children. It has been reported to occur in approximately one of 3,000 to 4,000 unvaccinated children during the COVID-19 waves dominated by variant Alpha of SARS-CoV-2. However, the incidences following SARS-CoV-2 infection with variant delta and omicron, as well as among vaccinated children and adolescents with SARS-CoV-2 is yet unexplored.

The investigators aim to estimate the incidence of MIS-C and in vaccinated and unvaccinated children and adolescents following variants delta and omicron, and other complications of SARS-CoV-2 including complication due to SARS-CoV-2 lock-down, based on a nationwide prospective population-based cohort study.

DETAILED DESCRIPTION:
AIM The project seeks to estimate the incidences of MIS-C in vaccinated and unvaccinated children and adolescents following variants delta and omicron, and other complications of SARS-CoV-2 including complication due to SARS-CoV-2 lock-down, .

HYPOTHESIS The incidences of MIS-C following SARS-CoV-2 variant delta and omicron are similar to the risk following variant alpha in unvaccinated children and adolescents, while the incidences among vaccinated children and adolescents are significantly lower. Further, severe complications to SARS-CoV-2, e.g. PVL producing S aur. infection is increased, as well as severe RSV-complication in older children in the post-COVID-lock down RSV epidemic

METHOD Prospective nationwide population-based cohort study of all individuals aged 0-17 years hospitalized due to MIS-C, or other complications to SARS-CoV-2 in the period August 15, 2021 to August 14, 2022. The setting is a multicenter study including all 18 Danish Pediatric Departments, providing 24 hours emergency service, and in- and out-patient treatment for all Danish inhabitants aged ≤ 17 years. As part of a pediatric nationwide COVID-19 research set-up, all 18 departments have a principal investigator responsible for prospective real-time data collection of patients with MIS-C and other complications to SARS-CoV-2, including complications secondary to the lock-down.

To calculate the incidence of MIS-C among Danish children and adolescents, the number of individuals who has tested positive for a SARS-CoV-2 infection in the period July 15 2021 to July 14 2022 will be attained from the National COVID-19-vaccine Database at the Statens Serum Institut. From the Statens Serum Institut and the Danish Microbiological Departments, the numbers bacterial infections including PVL-producing S aureus bacteremias and RSV infection will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* MIS-C according to criteria devised by the World Health Organization and Centers for Disease Control and Prevention (CDC)
* Invasive bacterial infections and viral infections secondary to SARS-CoV-2 or as consequence of SARS-CoV-2 lock down

Exclusion Criteria:

-

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children and adolescents in the whole population of Denmark
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-07-15 (Actual); Primary Completion 2024-07-14 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of MIS-C, invasive bacterial and viral infections | August to December 2021 (Delta); December 2021 to unknown (2022) (Omicron)

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen University Hospital Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Nygaard U, Hartling UB, Nielsen J, Vestergaard LS, Dungu KHS, Nielsen JSA, Sellmer A, Matthesen AT, Kristensen K, Holm M. Hospital admissions and need for mechanical ventilation in children with respiratory syncytial virus before and during the COVID-19 pandemic: a Danish nationwide cohort study. Lancet Child Adolesc Health. 2023 Mar;7(3):171-179. doi: 10.1016/S2352-4642(22)00371-6. Epub 2023 Jan 9. PMID 36634692
- [Derived] Nygaard U, Holm M, Hartling UB, Glenthoj J, Schmidt LS, Nordly SB, Matthesen AT, von Linstow ML, Espenhain L. Incidence and clinical phenotype of multisystem inflammatory syndrome in children after infection with the SARS-CoV-2 delta variant by vaccination status: a Danish nationwide prospective cohort study. Lancet Child Adolesc Health. 2022 Jul;6(7):459-465. doi: 10.1016/S2352-4642(22)00100-6. Epub 2022 May 6. PMID 35526537